CLINICAL TRIAL: NCT00548275
Title: Reducing Sex-Related HIV Risk Behaviors in Patients Receiving Treatment for Opioid Dependence
Acronym: Project RED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0609001848
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Opiate Dependence; HIV Infections
Keywords: Buprenorphine; Drug counseling; HIV risk reduction counseling; HIV Seronegativity; HIV risk behaviors
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Enhanced Sexual Risk Management (ESRM): Patients assigned to ESRM will attend 4 individual gender-specific interactive counseling sessions, once weekly over a four-week period. They will attend 2 sessions (20 minutes, weeks 2 and 3) followed by 2 sessions (40 minutes, weeks 4 and 5) that will be gender-specific to the patient and gender-matched with the study physicians (one female and one male) who will be trained in HIV testing and risk counseling. Sessions will include skill-building in condom use, safer sex negotiation, self-control of triggers and coping skills, didactic materials, and distribution of written material and address self-perception of risk, barriers to risk reduction, and negotiation of a risk-reduction plan.
  Interventions: Behavioral: Enhanced Sexual Risk Management
- 2 (Active Comparator): Standard Sexual Risk Management (SSRM): In SSRM, patients will attend two 10-minute gender non-specific individual educational sessions about HIV/AIDS provided by one of the study physicians who will be trained in HIV testing and risk counseling. Session 1 will coincide with the physician visit at the time of randomization. The patient will receive pre-test counseling at this time and undergo HIV antibody testing. Session 2 will take place 7 days later when the patient returns to receive their HIV test results and post-test counseling. In addition, subjects will receive didactic prevention messages about HIV relevant to their reported risks and will be asked if they have questions regarding this information.
  Interventions: Behavioral: Standard Sexual Risk Management

INTERVENTIONS:
Behavioral: Enhanced Sexual Risk Management — management of sexual risk
  Arms: 1
Behavioral: Standard Sexual Risk Management — management of sexual risk
  Arms: 2

SUMMARY:
The major goal is to determine in patients entering buprenorphine treatment, the prevalence of specific sex-related HIV risk behaviors, their physician's screening of these behaviors and to evaluate the impact of risk reduction counseling.

DETAILED DESCRIPTION:
The profile of opioid dependence is changing in the United States. According to the 2006 National Survey on Drug Use and Health (NSDUH), 3.7 million Americans had used heroin at least once in their lifetime and over half a million individuals had used heroin within the past year. Approximately 323,000 individuals met criteria for past-year heroin abuse or dependence. While these figures are concerning, the increasing prevalence of prescription opioid abuse and dependence is also worrisome. In 2006 12.6 million reported non-medical use of prescription opioids. Of these, 1.6 million met criteria for prescription opioid abuse or dependence. Sex-related HIV risk behaviors are prevalent amongst opioid dependent individuals with one study reporting unprotected intercourse within the prior 30 days in 75% of patients. Given that 79-85% of U.S. HIV/AIDS cases are secondary to sexual transmission, as non-injecting drug use increases, the relative contribution of sex-related HIV risk behaviors will increase as well. While drug treatment with methadone, and more recently buprenorphine (BUP), a new medication effective for the treatment of opioid dependence that can be prescribed by office-based physicians, has been shown to decrease drug-related HIV risk behaviors, my prior research demonstrates that BUP does not appear to impact as significantly on sex-related HIV risk behaviors. While the process of HIV risk behavior change begins with risk assessment, studies have shown that physicians, in general, frequently do not address risky behaviors with their patients. The current literature is lacking, however, with regards to the prevalence of specific high-risk sexual behaviors in patients enrolled in BUP treatment. Interventions specifically targeted at counseling for sex-related HIV risk behaviors delivered to patients receiving BUP treatment have not been refined. The proposed research will evaluate the prevalence of specific sex-related HIV risk behaviors in patients enrolled in office-based BUP treatment and the patients' perception of their providers' screening for these behaviors (Phase 1). These results will inform the conduct of a subsequent randomized clinical trial to evaluate the efficacy of a sex-related HIV risk reduction counseling intervention (Phase 2).

Phase 1. We hypothesize that sex-related HIV risk behaviors are prevalent in opioid dependent patients enrolled in BUP treatment and that patients will report that their providers fail to screen for these behaviors. The specific aims are to determine in patients entering BUP treatment: 1) the prevalence of specific sex-related HIV risk behaviors, and 2) by patient report, their provider's screening of these behaviors.

Phase 2. We hypothesize that in opioid dependent patients receiving office-based BUP, Enhanced Sexual Risk Management (ESRM) will be more effective in increasing specific safe sex practices compared with standard physician counseling, Standard Sexual Risk Management (SSRM) and that it will demonstrate cost-effectiveness overall when compared to SSRM. The specific aims of this randomized clinical trial are 1) to determine the efficacy of ESRM compared to SSRM, in individuals enrolled in BUP treatment and 2) To compare the cost-effectiveness of ESRM versus SSRM in individuals enrolled in BUP treatment. These interventions will be adapted from existing effective interventions evaluated in two recently conducted multi-site randomized clinical trials, the CDC-funded Project RESPECT and the NIMH-funded Project Light.20, 21

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting DSM-IV criteria for current opioid dependence
* HIV risk behaviors

Exclusion Criteria:

* current dependence on benzodiazepines or sedatives
* current suicide or homicide risk
* current psychotic disorder or untreated major depression
* inability to read or understand English
* unstable medical problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
proportion of condom use during acts of sexual intercourse | 3 months
number of unprotected vaginal/anal intercourse acts | 3 months
number of sexual partners | 3 months
recent diagnosis of an STD | 3 months

SECONDARY OUTCOMES:
buprenorphine treatment retention | 3 months
abstinence from illicit drug use | 3 months
health status | 3 months
patient and physician satisfaction | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E Sullivan, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Methadone Research Unit, The APT Foundation, Inc., New Haven, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut